CLINICAL TRIAL: NCT05270824
Title: Study Evaluating Neoadjuvant Immunotherapy Increasing CD8+ Cell Infiltration in Advance Gastric Adenocarcinoma : a Single Randomized Controlled Trial
Brief Title: Study Evaluating Neoadjuvant Immunotherapy Increasing CD8+ Cell Infiltration in Advance Gastric Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., chief physician, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUGES-025
Record Dates: First submitted 2022-02-22; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Advanced Gastric Carcinoma; CD8+ Tumor Infiltrating Lymphocytes; Neoadjuvant Immunotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radical surgery after neoadjuvant immunotherapy (albumin Paclitaxel + Seggio + PD-1 inhibitor) (Experimental): After randomization, patients received radical surgery after the neoadjuvant immunotherapy (albumin Paclitaxel + Seggio + PD-1 inhibitor)
  Interventions: Combination Product: radical surgery after neoadjuvant immunotherapy
- radical surgery after neoadjuvant chemotherapy (albumin Paclitaxel + Seggio) (Active Comparator): After randomization, patients received radical surgery after neoadjuvant chemotherapy (albumin Paclitaxel + Seggio)
  Interventions: Combination Product: radical surgery after neoadjuvant chemotherapy

INTERVENTIONS:
Combination Product: radical surgery after neoadjuvant immunotherapy — A total or distal gastrectomy with D2 lymph node dissection was done depending on the tumor location after neoadjuvant immunotherapy.
  Arms: radical surgery after neoadjuvant immunotherapy (albumin Paclitaxel + Seggio + PD-1 inhibitor)
Combination Product: radical surgery after neoadjuvant chemotherapy — A total or distal gastrectomy with D2 lymph node dissection was done depending on the tumor location after neoadjuvant immunotherapy.
  Arms: radical surgery after neoadjuvant chemotherapy (albumin Paclitaxel + Seggio)

SUMMARY:
Focusing on the clinical question of whether patients with advanced gastric cancer can benefit from immunotherapy, this project intends to detect the degree of CD8+ tumor-infiltrating lymphocyte infiltration in patients with advanced gastric cancer before and after receiving neoadjuvant combined immunotherapy and neoadjuvant therapy alone. To explore the evolving nature of tumor immune response before and after neoadjuvant therapy for gastric cancer, and quantitatively present it through chemical immunohistochemical techniques to achieve a more accurate diagnosis and treatment and improve the long-term efficacy of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 75 years
2. Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically ；
3. CT/MRI, PET-CT, or laparoscopic exploration should be performed before surgery to confirm the diagnosis of stage ≥cT2 or N+；
4. Patients who have not received other treatments such as surgery, radiotherapy, chemotherapy, targeted therapy or immunotherapy；
5. Performance status of 0 or 2 on Eastern Cooperative Oncology Group scale (ECOG)；
6. Estimated survival time was over 3 months；
7. No serious heart, lung and liver dysfunction; no jaundice and gastrointestinal obstruction; no acute infection;；
8. The major organs are functioning normally and meet the following criteria:

(1) Blood routine examination should meet the requirements (no blood transfusion within 14 days):

1. HB≥100g/L，
2. WBC≥3×109/L
3. ANC≥1.5×109/L，
4. PLT≥100×109/L； （2）Biochemical tests must meet the following criteria：

a. BIL <1.5×upper limit of normal (ULN)， b. ALT and AST<2.5ULN，GPT≤1.5×ULN； c. Cr≤1ULN，Ccr >60ml/min 9. Fertile women must have taken a pregnancy test (serum) within 7 days prior to enrollment with negative results and be willing to use an appropriate method of contraception during the trial period and 8 weeks after the last trial drug; For men, they should be surgically sterilized or agree to use the appropriate method of contraception during the trial period and 8 weeks after the last administration of the trial drug 10. Did not participate in other clinical studies before and during treatment 11. Subjects voluntarily joined the study and signed informed consent with good compliance and follow-up

Exclusion Criteria:

1. History of other malignant disease within past five years；
2. History of immunodeficiency, including HIV positive, or other acquired congenital immunodeficiency disease, or a history of organ transplantation and allogeneic bone marrow transplantation；
3. Contraindications to surgery and chemotherapy, or whose physical condition and organ function do not allow for major abdominal surgery
4. Distant metastases；
5. Accompanied by severe heart, lung, liver and kidney diseases; neurological and mental diseases; jaundice and accompanied by severe infection；
6. Women during pregnancy or breast-feeding；
7. Patients with high blood pressure that cannot be reduced to the normal range after antihypertensive drug treatment (systolic blood pressure>140 mmHg, diastolic blood pressure>90 mmHg);
8. Suffering from coronary heart disease of grade I or above, arrhythmia (including QTc interval prolongation > 450 ms in men and > 470 ms in women), and cardiac insufficiency;
9. Patients with a clear tendency to gastrointestinal bleeding, including the following conditions: patients with locally active ulcer lesions, fecal occult blood (++), and history of melena and hematemesis within 2 months; patients with abnormal coagulation function (INR> 1.5, APTT>1.5 ULN);
10. Patients with a history of cardiovascular and cerebrovascular diseases who are still taking oral thrombolytics or anticoagulants;
11. Patients with positive urine protein (urinary protein test 2+ or above, or 24-hour urine protein quantitative> 1.0g;
12. Multiple factors affect oral drugs (such as inability to swallow, persistent uncontrollable nausea and vomiting, chronic diarrhea and intestinal obstruction, etc.);
13. Those who have allergic reactions to the drugs in this study;
14. The researcher believes that it is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
The number of CD8+ tumor-infiltrating lymphocytes in tumor tissue and adjacent tissue before and after treatment | 6 months
  Changes in the number of CD8+ tumor-infiltrating lymphocytes in the tumor and adjacent tissues of the experimental group before and after the surgery compared with the control group.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 6 months
  Complete response (CR) + partial response (PR)
Disease-free survival (DFS) | 2 years
  Time from study entry to disease recurrence or patient death due to disease progression
Overall survival (OS) | 2 years
  Time from study entry to death from any cause.
Therapeutic drug safety | 6 months
  Adverse events (AEs), serious adverse events (SAEs), drug-related AEs, SAEs, and class-specific AEs (eg, hypertension, proteinuria, and hand-foot syndrome)
Surgical safety | 6 months
  R0 resection rate, operative mortality, surgical complications (bleeding, anastomotic leakage, incision infection), reoperation rate, hospital stay, etc.